CLINICAL TRIAL: NCT04061330
Title: Comparison of Low-dose Ketamine to Opioids in the Management of Acute Pain in Patients Presenting to the Emergency Department With Long Bone Fractures
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was terminated prior to enrollment due to lack of funding
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Paulina Sergot, Associate Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSC-MS-19-0580
Record Dates: First submitted 2019-08-15; First posted 2019-08-19 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: Pain, Acute
MeSH Terms: conditions — Acute Pain | interventions — Ketamine; Morphine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ketamine Group (Experimental)
  Interventions: Drug: Ketamine
- Opioid group (Active Comparator)
  Interventions: Drug: Morphine

INTERVENTIONS:
Drug: Ketamine — Initial bolus of ketamine 0.3 mg/kg IV (maximum 30 mg) followed by ketamine infusion of 0.25mg/kg/hr (maximum 25mg/kg/hr) for 6 hours or until patient leaves the emergency department (ED),whichever occurs first.
  Arms: Ketamine Group
Drug: Morphine — Bolus doses of morphine 0.1 mg/kg (maximum 8 mg) intravenously every 2 hours for 6 hours or until patient leaves the ED, whichever occurs first.
  Arms: Opioid group

SUMMARY:
The purpose of this study is to establish the feasibility of initiating a ketamine pain control protocol in the emergency department for the treatment of acute pain in patients with long bone fractures and to compare the efficacy of the ketamine pain protocol to bolus morphine for pain control in the first 6 hours of patient stay in the emergency department.

ELIGIBILITY:
Inclusion Criteria:

* patients presenting to the ED with long bone fracture, open or closed.Long bone fractures include:humerus, radius, ulna, femur, tibia, fibula.

Exclusion Criteria:

* Received morphine in the ED prior to enrollment
* Received ketamine any time prior to enrollment
* Glasgow Coma Scale(GCS) less than 15
* Transferred from other facility
* Other moderate to severe trauma injuries
* Contraindication to ketamine
* Cannot consent (no intubation, airway issues, hemodynamic instability)
* Prisoners
* Suspected and/or confirmed pregnancy

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2022-01-01 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinical pain as assessed by the Numerical pain rating score (NPRS) | baseline
  The NPRS total score ranges form 0-10,0 being no pain and 10 being worst possible pain.
Clinical pain as assessed by the Numerical pain rating score (NPRS) | 5 minutes after initial administration of drug
  The NPRS total score ranges form 0-10,0 being no pain and 10 being worst possible pain.
Clinical pain as assessed by the Numerical pain rating score (NPRS) | 10 minutes after initial administration of drug
  The NPRS total score ranges form 0-10,0 being no pain and 10 being worst possible pain.
Clinical pain as assessed by the Numerical pain rating score (NPRS) | 30 minutes after initial administration of drug
  The NPRS total score ranges form 0-10,0 being no pain and 10 being worst possible pain.
Clinical pain as assessed by the Numerical pain rating score (NPRS) | 60 minutes after initial administration of drug
  The NPRS total score ranges form 0-10,0 being no pain and 10 being worst possible pain.
Clinical pain as assessed by the Numerical pain rating score (NPRS) | 2 hours after initial administration of drug
  The NPRS total score ranges form 0-10,0 being no pain and 10 being worst possible pain.
Clinical pain as assessed by the Numerical pain rating score (NPRS) | 3 hours after initial administration of drug
  The NPRS total score ranges form 0-10,0 being no pain and 10 being worst possible pain.
Clinical pain as assessed by the Numerical pain rating score (NPRS) | 4 hours after initial administration of drug
  The NPRS total score ranges form 0-10,0 being no pain and 10 being worst possible pain.
Clinical pain as assessed by the Numerical pain rating score (NPRS) | 5 hours after initial administration of drug
  The NPRS total score ranges form 0-10,0 being no pain and 10 being worst possible pain.
Clinical pain as assessed by the Numerical pain rating score (NPRS) | 6 hours after initial administration of drug
  The NPRS total score ranges form 0-10,0 being no pain and 10 being worst possible pain.

SECONDARY OUTCOMES:
Number of hypoxic episodes as measured with a continuous pulse oximeter | 5 minutes after initial administration of drug
  Hypoxic episodes occur when peripheral capillary oxygen saturation (SPO2) is less than 90 percent as measured by a continuous pulse oximeter.
Number of hypoxic episodes as measured with a continuous pulse oximeter | 10 minutes after initial administration of drug
  Hypoxic episodes occur when peripheral capillary oxygen saturation (SPO2) is less than 90 percent as measured by a continuous pulse oximeter.
Number of hypoxic episodes as measured with a continuous pulse oximeter | 30 minutes after initial administration of drug
  Hypoxic episodes occur when peripheral capillary oxygen saturation (SPO2) is less than 90 percent as measured by a continuous pulse oximeter.
Number of hypoxic episodes as measured with a continuous pulse oximeter | 60 minutes after initial administration of drug
  Hypoxic episodes occur when peripheral capillary oxygen saturation (SPO2) is less than 90 percent as measured by a continuous pulse oximeter.
Number of hypoxic episodes as measured with a continuous pulse oximeter | 2 hours after initial administration of drug
  Hypoxic episodes occur when peripheral capillary oxygen saturation (SPO2) is less than 90 percent as measured by a continuous pulse oximeter.
Number of hypoxic episodes as measured with a continuous pulse oximeter | 3 hours after initial administration of drug
  Hypoxic episodes occur when peripheral capillary oxygen saturation (SPO2) is less than 90 percent as measured by a continuous pulse oximeter.
Number of hypoxic episodes as measured with a continuous pulse oximeter | 4 hours after initial administration of drug
  Hypoxic episodes occur when peripheral capillary oxygen saturation (SPO2) is less than 90 percent as measured by a continuous pulse oximeter.
Number of hypoxic episodes as measured with a continuous pulse oximeter | 5 hours after initial administration of drug
  Hypoxic episodes occur when peripheral capillary oxygen saturation (SPO2) is less than 90 percent as measured by a continuous pulse oximeter.
Number of hypoxic episodes as measured with a continuous pulse oximeter | 6 hours after initial administration of drug
  Hypoxic episodes occur when peripheral capillary oxygen saturation (SPO2) is less than 90 percent as measured by a continuous pulse oximeter.
Number of hypotension episodes | 5 minutes after initial administration of drug
  Hypotension occurs when systolic blood pressure (SBP) is less than 100mmHg
Number of hypotension episodes | 10 minutes after initial administration of drug
  Hypotension occurs when systolic blood pressure (SBP) is less than 100mmHg
Number of hypotension episodes | 30 minutes after initial administration of drug
  Hypotension occurs when systolic blood pressure (SBP) is less than 100mmHg
Number of hypotension episodes | 60 minutes after initial administration of drug
  Hypotension occurs when systolic blood pressure (SBP) is less than 100mmHg
Number of hypotension episodes | 2 hours after initial administration of drug
  Hypotension occurs when systolic blood pressure (SBP) is less than 100mmHg
Number of hypotension episodes | 3 hours after initial administration of drug
  Hypotension occurs when systolic blood pressure (SBP) is less than 100mmHg
Number of hypotension episodes | 4 hours after initial administration of drug
  Hypotension occurs when systolic blood pressure (SBP) is less than 100mmHg
Number of hypotension episodes | 5 hours after initial administration of drug
  Hypotension occurs when systolic blood pressure (SBP) is less than 100mmHg
Number of hypotension episodes | 6 hours after initial administration of drug
  Hypotension occurs when systolic blood pressure (SBP) is less than 100mmHg
Score on Richmond Agitation-Sedation Scale (RASS) | 5 minutes after initial administration of drug
  The RASS is a 10-point scale ranging from +4 to -5, with four levels of anxiety or agitation (+4 to +1), one level denoting a calm and alert state (0), and 5 levels of sedation (-1 to -5). +4 represents a very combative, violent patient, and on the other extreme -5 represents a patient who is unarousable, with no response to voice or physical stimulation.
Score on Richmond Agitation-Sedation Scale (RASS) | 10 minutes after initial administration of drug
  The RASS is a 10-point scale ranging from +4 to -5, with four levels of anxiety or agitation (+4 to +1), one level denoting a calm and alert state (0), and 5 levels of sedation (-1 to -5). +4 represents a very combative, violent patient, and on the other extreme -5 represents a patient who is unarousable, with no response to voice or physical stimulation.
Score on Richmond Agitation-Sedation Scale (RASS) | 30 minutes after initial administration of drug
  The RASS is a 10-point scale ranging from +4 to -5, with four levels of anxiety or agitation (+4 to +1), one level denoting a calm and alert state (0), and 5 levels of sedation (-1 to -5). +4 represents a very combative, violent patient, and on the other extreme -5 represents a patient who is unarousable, with no response to voice or physical stimulation.
Score on Richmond Agitation-Sedation Scale (RASS) | 60 minutes after initial administration of drug
  The RASS is a 10-point scale ranging from +4 to -5, with four levels of anxiety or agitation (+4 to +1), one level denoting a calm and alert state (0), and 5 levels of sedation (-1 to -5). +4 represents a very combative, violent patient, and on the other extreme -5 represents a patient who is unarousable, with no response to voice or physical stimulation.
Score on Richmond Agitation-Sedation Scale (RASS) | 2 hours after initial administration of drug
  The RASS is a 10-point scale ranging from +4 to -5, with four levels of anxiety or agitation (+4 to +1), one level denoting a calm and alert state (0), and 5 levels of sedation (-1 to -5). +4 represents a very combative, violent patient, and on the other extreme -5 represents a patient who is unarousable, with no response to voice or physical stimulation.
Score on Richmond Agitation-Sedation Scale (RASS) | 3 hours after initial administration of drug
  The RASS is a 10-point scale ranging from +4 to -5, with four levels of anxiety or agitation (+4 to +1), one level denoting a calm and alert state (0), and 5 levels of sedation (-1 to -5). +4 represents a very combative, violent patient, and on the other extreme -5 represents a patient who is unarousable, with no response to voice or physical stimulation.
Score on Richmond Agitation-Sedation Scale (RASS) | 4 hours after initial administration of drug
  The RASS is a 10-point scale ranging from +4 to -5, with four levels of anxiety or agitation (+4 to +1), one level denoting a calm and alert state (0), and 5 levels of sedation (-1 to -5). +4 represents a very combative, violent patient, and on the other extreme -5 represents a patient who is unarousable, with no response to voice or physical stimulation.
Score on Richmond Agitation-Sedation Scale (RASS) | 5 hours after initial administration of drug
  The RASS is a 10-point scale ranging from +4 to -5, with four levels of anxiety or agitation (+4 to +1), one level denoting a calm and alert state (0), and 5 levels of sedation (-1 to -5). +4 represents a very combative, violent patient, and on the other extreme -5 represents a patient who is unarousable, with no response to voice or physical stimulation.
Score on Richmond Agitation-Sedation Scale (RASS) | 6 hours after initial administration of drug
  The RASS is a 10-point scale ranging from +4 to -5, with four levels of anxiety or agitation (+4 to +1), one level denoting a calm and alert state (0), and 5 levels of sedation (-1 to -5). +4 represents a very combative, violent patient, and on the other extreme -5 represents a patient who is unarousable, with no response to voice or physical stimulation.
Number of participants with need for rescue opioid therapy | from time of initial administration of drug to end of treatment (about 6 hours after initial administration of drug)
Number of participants with need for rescue benzodiazepine therapy in ketamine group for emergence phenomenon and dysphoria | from time of initial administration of drug to end of treatment (about 6 hours after initial administration of drug)
Number of participants with Adverse reactions | from time of initial administration of drug to end of treatment (about 6 hours after initial administration of drug)
Patient satisfaction with analgesia | end of treatment (about 6 hours after initial administration of drug)
  Patient satisfaction will be measured on a 5 point scale, with 1 being very unsatisfied and 5 being very satisfied.
Physician satisfaction with analgesia | end of treatment (about 6 hours after initial administration of drug)
  Physician satisfaction will be measured on a 5 point scale, with 1 being very unsatisfied and 5 being very satisfied.
Nursing satisfaction with analgesia | end of treatment (about 6 hours after initial administration of drug)
  Nursing satisfaction will be measured on a 5 point scale, with 1 being very unsatisfied and 5 being very satisfied.

CONTACTS AND LOCATIONS:
Overall Officials: Paulina Sergot, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No